CLINICAL TRIAL: NCT07162506
Title: Definitive Concurrent Chemoradiotherapy Versus Surgery in Patients With Locally Advanced Resectable Esophageal Squamous Cell Carcinoma (ESCC) Who Achieve Complete or Partial Response After Neoadjuvant Camrelizumab Combined With Chemotherapy: A Two-arm Phase II Clinical Study (SORT Trial)
Brief Title: DCRT vs. Surgery in Resectable ESCC Patient Achiving cCR/PR After nCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Wencheng Zhang, Associated Prof. in the department of radiation oncology, Tianjin Medical University Cancer Institute and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20250845A
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Radical esophagectomy + mediastinal lymph node dissection
  Interventions: Procedure: Surgery
- DCRT (Experimental): Definitive concurrent chemoradiotherapy (radiotherapy: 50.4 Gy/28f; chemotherapy: nab-paclitaxel 175mg/m² + carboplatin AUC=5, q21d for 2 cycles)
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Procedure: Surgery — Radical esophagectomy + mediastinal lymph node dissection
  Arms: Surgery
Radiation: Radiotherapy — Radiotherapy: 50.4 Gy/28f
  Arms: DCRT
Drug: Chemotherapy — Chemotherapy: nab-paclitaxel 175mg/m² + carboplatin AUC=5, q21d for 2 cycles
  Arms: DCRT

SUMMARY:
This is a single-center, Phase II clinical study aiming to evaluate the efficacy, safety, and organ preservation feasibility of definitive concurrent chemoradiotherapy versus surgery in patients with locally advanced resectable esophageal squamous cell carcinoma (ESCC) who achieve clinical complete response/partial response (cCR/PR) after neoadjuvant camrelizumab combined with chemotherapy.

A total of 120 eligible subjects will be enrolled. Patients with cCR/PR after 2 cycles of induction chemoimmunotherapy (camrelizumab + nab-paclitaxel + carboplatin) will be grouped based on personal willing: the control group (n=60) will receive radical esophagectomy + mediastinal lymph node dissection; the experimental group (n=60) will receive definitive concurrent chemoradiotherapy (radiotherapy: 50.4 Gy/28f; chemotherapy: nab-paclitaxel 175mg/m² + carboplatin AUC=5, q21d for 2 cycles). All the patients will receive camrelizumab maintenance therapy (200mg q21d) up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate, cooperated with follow-up visits.
2. Aged 18 - 75 years (inclusive), male or female.
3. Histologically confirmed locally advanced resectable ESCC, clinically staged as Stage II - IVa (cT1N1-3M0, cT2-4aN0-3M0 before treatment; 8th AJCC), and achieve cCR/PR after 2 cycles of camrelizumab combined with nab-paclitaxel and carboplatin.
4. Presence of measurable and/or non-measurable lesions as defined by Japanese Classification of Esophageal Cancer (12th Edition);
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Estimated survival time ≥ 3 months.
7. The function of major organs meets the following requirements:

   1. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L;
   2. Platelets ≥ 80×10^9/L;
   3. Hemoglobin ≥ 9g/dL;
   4. Serum albumin ≥ 2.8g/dL;
   5. Total bilirubin ≤ 1.5 × ULN, ALT, AST and/or ALP ≤ 2.5 × ULN;
   6. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60mL/min;
   7. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5× ULN (subjects on stable doses of anticoagulation therapy, such as low molecular weight heparin or warfarin, and with INR within the expected therapeutic range of the anticoagulant can be screened);
8. Patients of childbearing potential must use a medically approved contraceptive method (such as intrauterine device, contraceptive pills, or condoms) during the study treatment period and within 6 months after the end of the study treatment; serum Human Chorionic Gonadotropin (HCG) or urine HCG test must be negative within 72 hours before study enrollment; and must not be breastfeeding.

Exclusion Criteria:

1. Surgery for esophageal cancer;
2. Esophageal fistulae due to infiltration of the primary tumor；
3. Risk of gastrointestinal bleeding, esophageal fistula or esophageal perforation;
4. Poor nutritional status, weight loss of ≥10% in the previous 2 months, with no significant improvement after nutritional intervention;
5. Major surgery or severe trauma within 4 weeks prior to first use of study drug;
6. Uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
7. Received or receiving any of the following treatments in the past:

   1. Anti-PD-1 (except for camrelizumab) or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy or targeted therapy;
   2. Participation in a study of an investigational agent or device within 4 weeks before the first dose of study treatment;
   3. Systemic treatment with corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressive agents is required for 2 weeks before the first dose of study treatment (except for the use of corticosteroids for local inflammation of the esophagus and for the prevention of allergy and nausea and vomiting). Other special circumstances need to be communicated to the sponsor. Inhaled or topical steroids and adrenocorticotropic hormone replacement at doses >10mg/day prednisone efficacy dose are permitted if the patient does not have active autoimmune disease;
   4. Received an anti-tumour vaccine or received a live vaccine within 4 weeks before the first dose of study treatment;
8. Any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Except for patients with vitiligo or those who had asthma or allergies in childhood but did not need any intervention as adults; patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes mellitus treated with stable doses of insulin may be included;
9. Diagnosis of immunodeficiency, including positive HIV test, other acquired/congenital immunodeficiency diseases, organ transplantation and allogeneic bone marrow transplantation;
10. Diagnosis of uncontrolled cardiac clinical symptoms or disease such as: a. NYHA II or above heart failure; b. unstable angina; c. myocardial infarction within 1 year; d. clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
11. Severe infections (CTCAE > grade 2), such as severe pneumonia requiring hospitalisation, bacteraemia, infectious co-morbidities, etc., within 4 weeks before the first use of study treatment; Baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks before the first use of study treatment, except for prophylactic antibiotic use;
12. History of interstitial lung disease or non-infectious pneumonia, or pulmonary insufficiency ≥ grade 3 as confirmed by pulmonary function tests;
13. Active tuberculosis infection detected by history or CT examination, or history of active tuberculosis infection within 1 year before enrollment or more than 1 year previously without regular treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection);
15. Presence of abnormal sodium, potassium, and calcium laboratory test values greater than grade 1 within 2 weeks prior to enrollment that do not improve with treatment;
16. Known hypersensitivity to large protein preparations, or to any of the components of camrelizumab, or anaphylaxis, hypersensitivity, or contraindication to paclitaxel or carboplatin or to any of the components used within their preparations;
17. Previously diagnosed with any other malignancy before the first use of the investigational drug, except for malignancies with low risk of metastasis and death (5-year survival rate>90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
18. As judged by the investigator, the subject has other factors that may lead to forced termination of the study midway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
DFS | up to 3 years
  Disease-Free Survival

SECONDARY OUTCOMES:
OS | up to 3 years
  Overall Survival
LRR | up to 3 years
  locoregional disease recurrence
R0 resection | up to 3 years
  Surgical and pathological outcome
AEs | up to 3 years
  Adverse Events
QoL | up to 3 years
  Quality of Life score
PG - SGA | up to 3 years
  Patient - Generated Subjective Global Assessment Scale
SSA | up to 3 years
  Standardized Swallowing Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Zhang, M.D., Principal Investigator — Tianjin Cancer Hospital; Xiaofeng Duan, M.D., Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No